CLINICAL TRIAL: NCT05789043
Title: Camrelizumab in Combination With Apatinib and Temozolomide as First-line Treatment in Advanced Acral Melanoma: a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Camrelizumab in Combination With Apatinib and Temozolomide as First-line Treatment in Advanced Acral Melanoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Chief physician, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-MM-III-004
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Acral Melanoma
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Three-drug arm (Experimental)
  Interventions: Drug: camrelizumab+apatinib+TMZ
- Two-drug arm (Active Comparator)
  Interventions: Drug: camrelizumab+apatinib
- single-drug arm (Active Comparator)
  Interventions: Drug: camrelizumab

INTERVENTIONS:
Drug: camrelizumab+apatinib+TMZ — camrelizumab 200mg，q2w+apatinib 250mg，qd+TMZ 200mg/m2，day1-5/28
  Arms: Three-drug arm
Drug: camrelizumab+apatinib — camrelizumab 200mg，q2w+apatinib 250mg qd
  Arms: Two-drug arm
Drug: camrelizumab — camrelizumab 200mg，q2w
  Arms: single-drug arm

SUMMARY:
It is a RCT aimed to evaluate the Progression Free Survival of Camrelizumab combined with apatinib and temozolomide as First Line Therapy in Advanced Acral Melanoma.

ELIGIBILITY:
Inclusion Criteria:

* age:≥18 years, male or female.
* Histopathologically confirmed recurrence, inoperable resection or metastatic acral melanoma (stage III/IV).
* Has not received any systematic anti-tumor drug treatment.
* Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
* ECOG 0-1.
* Adequate organ function.
* Life expectancy of greater than 12 weeks.
* Patient has given written informed consent.

Exclusion Criteria:

* Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
* Known history of hypersensitivity to macromolecular protein preparation or any components of the drug formulation.
* Subjects before or at the same time with other malignant tumors (except which has cured skin basal cell carcinoma and cervical carcinoma in situ);
* Subjects with any active autoimmune disease or history of autoimmune disease Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
* Received a live vaccine within 4 weeks before the first dose of study medication.
* Pregnancy or breast feeding.
* Decision of unsuitableness by principal investigator or physician-in charge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival, PFS | Within 2 years
  PFS was defined as the time from randomization to progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival ,OS | Within 2 years
  OS will be defined as the time from randomization to death due to any cause.
ORR | Within 2 years
  The objective response rate will be assessed by RECIST 1.1
DCR | Within 2 years
  The disease control rate will be assessed by RECIST 1.1
Adverse Events (AEs) | Within 2 years
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily had to have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Dr, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China